CLINICAL TRIAL: NCT04993885
Title: Efficacy and Safety of Avatrombopag in the Treatment of Adult Immune Thrombocytopenia With Autoantibodies Fail to Eltrombopag or Herombopag Treatment: a Single-center, Prospective, One-arm Clinical Trial
Brief Title: Avatrombopag in the Treatment of Adult Immune Thrombocytopenia With Autoantibodies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2021033
Record Dates: First submitted 2021-08-03; First posted 2021-08-06 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Immune Thrombocytopenia; Autoantibodies; Evan Syndrome; Connective Tissue Diseases
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Evans Syndrome; Connective Tissue Diseases | interventions — avatrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Fifty-two subjects will be enrolled with the indicated treatment dose of avatrombopag
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — The subjects will receive avatrombopag treatment with an initial dose of 40mg once a day. Platelet counts will be obtained weekly during the first 4 weeks and then every 2 weeks until week 12 after treatment. The dose adjustment range is 20 mg per week to 40 mg per day to maintain the platelet level between 30×10^9/L and 200×10^9/L. If the platelet count does not reach to 30×10^9/L after taking avatrombopag 40mg once a day for 4 consecutive weeks, the treatment will be stopped.

SUMMARY:
This prospective, open-label, single-center, one-arm clinical trial aims at evaluating the efficacy and safety of avatrombopag in Chinese adult Immune Thrombocytopenia (ITP) patients with autoantibodies fail (due to intolerance or resistance) to eltrombopag or herombopag treatment.

DETAILED DESCRIPTION:
This prospective, open-label, single-center, one-arm clinical trial aims at evaluating the efficacy and safety of avatrombopag in Chinese adult ITP patients with autoantibodies fail (due to intolerance or resistance) to eltrombopag or herombopag treatment.

The subjects include ITP secondary to connective tissue diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome and rheumatoid arthritis), primary ITP with positive antinuclear antibody but not up to the diagnostic criteria of connective tissue diseases, primary Evans syndrome, Evans syndrome secondary to connective tissue diseases, and primary ITP with positive Coomb's test but not up to the diagnostic criteria of Evans syndrome.

Fifty-two eligible subjects will be enrolled in this study. The dose will be adjusted according to the platelet count during the period from week 1 to week 12.

ELIGIBILITY:
Inclusion Criteria:

* The patients have provided written informed consent prior to enrollment.
* Men and women greater than or equal to 18 years of age.
* Diagnosed as ITP secondary to connective tissue diseases (including but not limited to systemic lupus erythematosus, Sjogren's syndrome and rheumatoid arthritis), primary ITP with positive antinuclear antibody but not up to the diagnostic criteria of connective tissue diseases, primary Evans syndrome, Evans syndrome secondary to connective tissue diseases, and primary ITP with positive Coomb's test but not up to the diagnostic criteria of Evans syndrome.
* Platelet count<30 ×10^9/L at screening.
* Patients who have previously failed to receive Eltrombopag or Herombopag [poor efficacy (Eltrombopag 75 mg/d or Herombopag 7.5 mg/D, at least 4 weeks), or the efficacy cannot be maintained], or who have contraindications, can not tolerate or refuse Eltrombopag or Herombopag treatment.
* Treatment for ITP (including but not limited to glucocorticoids, recombinant human thrombopoietin, and other thrombopoietin receptor agonists other than Avatrombopag) must be completed before enrollment, or the dose must be stable or in a phase of reduction within 2 weeks before enrollment.
* Effective contraceptive measures will be taken during the clinical trial.

Exclusion Criteria:

* Patients with active thyroid disease requiring treatment.
* Patients with any prior history of arterial or venous thrombosis within 3 months, and with any of the following risk factors: cancer, Factor V Leiden, ATIII deficiency, or patients who are using anticoagulants or antiplatelet drugs at the beginning of screening.
* Those who had received rituximab within 3 months.
* Patients who had failed to respond to the previous use of Avatrombopag (40mg once a day for more than 4 weeks).
* Subjects known to be allergic to Avatrombopag or any of its excipients.
* Patients who had received splenectomy within 3 months or have splenectomy plan within 3 months.
* Patients with lupus encephalopathy or lupus nephritis.
* Patients with cataract.
* Patients with infectious fever (including but not limited to pulmonary infection) within 1 month or with active infection during screening.
* Existing hepatitis B virus, hepatitis C virus replication or HIV infection.
* Severe liver dysfunction (alanine aminotransferase or glutamic oxaloacetic transaminase > 3×ULN).
* Patients with severe cardiac or pulmonary dysfunction.
* Severe renal damage (creatinine clearance < 30 ml/min).
* There are surgical planners during the study.
* History of psychiatric disorder.
* Pregnant or lactating women or those planning to be pregnant during the trial.
* Patients with a history of drug/alcohol abuse (within 2 years before the study).
* Patients that had participated in other experimental researches within one month before enrollment.
* Any other circumstances that the investigator considers that the patient is not suitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Percentage of participants achieving a platelet count >=30×10^9/L and at least doubling of the baseline count within 12 weeks of treatment.

SECONDARY OUTCOMES:
Platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Proportion of subjects who achieve response (R) within 1, 2, 4 and 8 weeks of treatment.
Platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Proportion of subjects who achieve complete response (CR) within 4, 8 and 12 weeks of treatment.
Duration of platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Proportion of subjects with a platelet count >=30×10^9/L for at least 4 consecutive weeks during the 12 week treatment period without remedial treatment.
Platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Percentage of participants achieving a platelet count >=50×10^9/L within 12 weeks of treatment.
Time to platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Time to response is defined as time from the start of treatment to the first time of achieving a platelet count >= 30×10^9/L and at least doubling of the baseline count during the whole 12 weeks.
Duration of platelet response | From the start of study treatment (Day 1) up to the end of week 12.
  Total duration of time a participant with a response of R.
Proportion of patients receiving remedial treatment. | From the start of study treatment (Day 1) up to the end of week 12.
  Proportion of patients receiving remedial treatment.
Bleeding score | From the start of study treatment (Day 1) up to the end of week 12.
  The incidence and grade of bleeding symptoms according to the World Health Organization Bleeding Scale.
Changes of disease activity index in patients with systemic lupus erythematosus | From the start of study treatment (Day 1) up to the end of week 12.
  The proportion of subjects with improvement of disease activity index in patients with systemic lupus erythematosus according to the SLEDAI standard.
The improvement of symptoms | From the start of study treatment (Day 1) up to the end of week 12.
  The proportion of subjects with improvement of symptoms including skin symptom, joint pain, dry mouth and dry eyes.
Improvement in immune indexes | From the start of study treatment (Day 1) up to the end of week 12.
  The proportion of subjects with improvement immune indexes including antinuclear antibody, extractable nuclear antigens spectrum and Coomb's test.
Discontinuation rate of glucocorticoids | From the start of study treatment (Day 1) up to the end of week 12.
  The proportion of subjects with discontinuation use of glucocorticoids.
Functional assessment of chronic illness therapy-fatigue | From the start of study treatment (Day 1) up to the end of week 12.
  In all participants, functional assessment of chronic illness therapy-fatigue questionnaire will be used to assess the health related quality of life before and after treatment.
ITP-Patient Assessment Questionnaire | From the start of study treatment (Day 1) up to the end of week 12.
  In all participants, ITP-Patient Assessment Questionnaire will be used to assess the health related quality of life before and after treatment.

OTHER OUTCOMES:
Incidence of Toxicity | From the start of study treatment (Day 1) up to the end of week 12.
  The proportion of subjects with specific pre-defined toxicity, including headache, fever, nausea and abdominal pain, and unpredictable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, M.D., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China